CLINICAL TRIAL: NCT02911779
Title: The Optimal Angle of Mediolateral Episiotomy at Crowning of the Head During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Shimon Ginath, Medical Doctor OBGYN, Wolfson Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0181-11-WOMC
Record Dates: First submitted 2016-09-18; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Labor, Obstetric; Episiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- change of medilateral angle line (Other): change of medilateral angle line during crowning of the head
  Interventions: Procedure: change of medilateral angle line during crowning of the head

INTERVENTIONS:
Procedure: change of medilateral angle line during crowning of the head — change of medilateral angle line during crowning of the head

SUMMARY:
In order to determine the optimal angle to perform an episiotomy, the investigators assessed the angle of marked episiotomy lines at the first stage of labor and at the time of crowning of the head.

Incision lines for mediolateral episiotomy were pre-marked on the perineal skin at 30°, 45°, and 60° angles from the midline, at the first stage of labor, in women with singleton pregnancies. The angles of the marked lines were measured again at crowning of the head. Mediolateral episiotomy was performed only for obstetric indications.

ELIGIBILITY:
Inclusion Criteria:

* women during labor above 37 weeks, Occiput presentation

Exclusion Criteria:

* cesarean section, vacuum or forceps deliver, breech deliver, below 37 weeks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change of medilateral angle line during crowning of the head | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No